CLINICAL TRIAL: NCT05080842
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-Tumor Activity of AC682 in Patients With Estrogen Receptor Positive/Human Epidermal Growth Factor Receptor 2 Negative (ER+/HER2-) Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of AC682 for the Treatment of Locally Advanced or Metastatic ER+ Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Voluntarily terminate the study since the sponsor's development strategy was adjusted.
Sponsor: Accutar Biotechnology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC682-001
Record Dates: First submitted 2021-09-22; First posted 2021-10-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Estrogen receptor positive; ER positive; ER+; Human epidermal growth factor receptor 2 negative; HER2 negative; HER2-; AC682; Breast cancer; Phase I
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AC682 (Experimental): This arm will evaluate AC682 monotherapy administered in 28-day cycles. Up to 30 participants will participate in this dose escalation arm.
  Interventions: Drug: AC682

INTERVENTIONS:
Drug: AC682 — Participants will receive AC682 by mouth daily in 28-day cycles.

SUMMARY:
This clinical trial is evaluating a drug called AC682 in participants with estrogen receptor positive/human epidermal growth factor 2 negative (ER+/HER2-) locally advanced or metastatic breast cancer. The main goals of this study are to:

* Identify the recommended dose of AC682 that can be given safely to participants
* To evaluate the side effects of AC682
* To evaluate pharmacokinetics of AC682
* To evaluate the effectiveness of AC682

DETAILED DESCRIPTION:
This is a Phase I, first in human, open-label dose-escalation study of AC682, an orally available estrogen receptor degrader, given as a single agent.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form (ICF)
* Patients must be ≥18 years-of-age at the time of signing of the ICF
* Female patients must be postmenopausal
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Histologically and/or cytologically confirmed advanced estrogen receptor positive (ER+) human epidermal growth factor 2 negative (HER2-) breast cancer
* Patients with life expectancy ≥3 months
* Patients who have adequate organ functions at baseline
* At least 1 measurable lesion that meets the definition in Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 or at least 1 non-target lesion is required.

Exclusion Criteria:

* Treatment with any of the following: systemic anti-cancer chemotherapy, biologic, or hormonal agent from a previous treatment regimen or clinical study within 4 weeks prior to the first dose of AC682; systemic small molecules from a previous treatment regimen or clinical study within 14 days or 5 half-lives (whichever is longer) prior to the first dose of AC682 (at least 10 days must have elapsed between the last dose of such agent and the first dose of study drug)
* Radiation therapy such as wide-field radiotherapy administered ≤28 days of first dose of AC682
* Major surgery (excluding placement of vascular access) within 4 weeks of first dose of AC682
* Known symptomatic brain metastases requiring the use of steroids
* Any condition that impairs a patient's ability to swallow whole pills. Impairment of gastrointestinal function (GI) or GI disease or other condition at baseline that will interfere significantly with the absorption, distribution, or metabolism of AC682.
* Use of prophylactic growth factors and blood transfusions ≤14 days prior to the first dose of AC682 and during dose limiting toxicity observation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | 28 days (Cycle 1)
Incidence of treatment-emergent adverse events (TEAEs), and clinically significant grade 3 or higher laboratory abnormalities following administration of AC682 | Through study completion, approximately 18 months
  Adverse events will be graded according to NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Objective response rate (ORR) as a measure of anti-tumor activity | Through study completion, approximately 18 months
Clinical benefit rate (CBR) as a measure of anti-tumor activity | Through study completion, approximately 18 months
Duration of response (DOR) as a measure of anti-tumor activity | Through study completion, approximately 18 months
Disease control rate (DCR) as a measure of anti-tumor activity | Through study completion, approximately 18 months
Progression free survival (PFS) as a measure of anti-tumor activity | Through study completion, approximately 18 months
Pharmacokinetic Analysis: area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC(0-inf)) | Through study completion, approximately 18 months
Pharmacokinetic Analysis: area under the concentration-time curve over the dosing interval (AUC(0-tau)) | Through study completion, approximately 18 months
Pharmacokinetic Analysis: maximum plasma concentration (Cmax) | Through study completion, approximately 18 months
Pharmacokinetic Analysis: time to maximum plasma concentration (tmax) | Through study completion, approximately 18 months
Pharmacokinetic Analysis: terminal elimination half life (t1/2) | Through study completion, approximately 18 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Site 01, Denver, Colorado
  - Site 04, Orlando, Florida
  - Site 02, Sarasota, Florida
  - Site 03, Nashville, Tennessee
  - Site 05, Houston, Texas

IPD SHARING:
Plan to Share IPD: No